CLINICAL TRIAL: NCT05070637
Title: No-touch Radical Nephrectomy Technique Reduces Circulating Tumor Cell Release in Renal Cell Carcinoma Patients - a Randomized Controlled Trial
Brief Title: Circulating Tumor Cell Reducing No-touch Nephrectomy
Acronym: CITO-CERENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Collaborators: Instituto de Medicina Molecular João Lobo Antunes (Other); Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Tito Palmela Leitão, MD, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2021-09-26; First posted 2021-10-07 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Renal Cell Carcinoma; Circulating Tumor Cell
Keywords: circulating tumor cell; renal cell carcinoma; radical nephrectomy; no-touch nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplastic Cells, Circulating

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No-touch laparoscopic radical nephrectomy (Experimental): Group A patients will undergo a no-touch laparoscopic radical nephrectomy, with the dissection being done through the Gerota's fascia plane until exposure of the corresponding great vessel (vena cava on the right side, and aorta on the left side) is obtained. The renal pedicle will be directly isolated, and ligated using Weck® clips with no kidney manipulation.
  Interventions: Procedure: No-touch laparoscopic radical nephrectomy
- Conventional laparoscopic radical nephrectomy (Active Comparator): Group B patients will undergo a conventional laparoscopic radical nephrectomy approach, starting with opening of the Gerota's fascia, identification of the ureter, traction on the peri-renal fat below the ureter while dissecting cephalad until the renal pedicle is reached. The renal pedicle will then be isolated while maintaining traction on the kidney, and peri-renal fat, and ligated using Weck® clips.
  Interventions: Procedure: Conventional laparoscopic radical nephrectomy
- Laparoscopic total nephrectomy control arm (Other): Control arm in which a laparoscopic total nephrectomy will be performed in patients with hypo-functioning kidneys, and no renal cell carcinoma.
  Interventions: Procedure: Laparoscopic total nephrectomy control arm

INTERVENTIONS:
Procedure: No-touch laparoscopic radical nephrectomy — We aim to determine if a laparoscopic no-touch nephrectomy with an early renal pedicle ligation can decrease CTC release during surgery.
  Arms: No-touch laparoscopic radical nephrectomy
Procedure: Conventional laparoscopic radical nephrectomy — Conventional laparoscopic radical nephrectomy, which implies manipulation of the kidney, opening of the Gerota's fascia, and manipulation of peri-nephric fat during dissection, and renal pedicle isolation.
  Arms: Conventional laparoscopic radical nephrectomy
Procedure: Laparoscopic total nephrectomy control arm — Control arm in which a laparoscopic total nephrectomy will be performed in non-cancer patients.
  Arms: Laparoscopic total nephrectomy control arm

SUMMARY:
This study will study circulating tumor cell (CTC) release during laparoscopic radical nephrectomy (LRN) for RCC. The main objective is to determine if CTC release can be reduced during RN by using a no-touch technique, with an early renal pedicle ligation. The investigators also aim to describe the CTC profile in terms of CTC count (CTCn), epithelial/mesenchymal status, and CTC cellular features in renal cell carcinoma (RCC) patients, stratified by "primary tumor, regional nodes, metastasis" (TNM) staging, histological subtype, and other clinical and radiological features.

Patients undergoing RN will enter a two-arm prospective single-center randomized controlled trial (RCT), comparing a no-touch RN technique, with direct pedicle ligation (Group A) vs. the more conventional approach of kidney traction and manipulation to reach the renal pedicle before its ligation (Group B).

A microfluidic size-based CTC isolation device will be used to capture and count CTCs from peripheral blood samples of these patients. CTCs will be identified by staining with antibodies to cytokeratin 8/18, vimentin, 4',6-diamidino-2-phenylindole (DAPI), and cluster of differentiation antigen 45 (CD45).

CTC release will be correlated with the disease-free survival (DFS), and overall survival (OS). The investigators will determine if CTC reducing no-touch radical nephrectomy technique improves these hard outcomes.

DETAILED DESCRIPTION:
This study will study CTC profile in RCC, and their release into the blood circulation during LRN.

Included patients will be referred to the Renal Cancer Unit of the North Lisbon University Hospital Center (CHLUN) Urology Department with the diagnosis of a renal mass eligible for a LRN. Patients will have their diagnosis confirmed, be appropriately staged, and their management options will be decided after a shared and informed decision process in light of the current European Association of Urology (EAU) Guidelines on RCC. Patients < 18 years old and pregnant women will be excluded. Patients will be adequately informed of the study protocol, and will sign a specific informed consent.

Patients undergoing LRN will enter a two-arm prospective single-center randomized controlled trial, comparing a no-touch technique, with direct pedicle ligation (Group A) vs. the conventional dissection, and ligation of the renal pedicle with kidney traction (Group B). A peripheral blood sample will be collected at arrival to the operating room. After that, Group A patients will undergo a no-touch RN, with the dissection being done through the Gerota's fascia plane until exposure of the corresponding great vessel (vena cava on the right side, and aorta on the left side) is obtained. The renal pedicle will be directly isolated, and ligated using Weck® clips with no kidney manipulation. Group B patients will undergo a more conventional approach, starting with opening of the Gerota's fascia, identification of the ureter, traction on the peri-renal fat below the ureter while dissecting cephalad until the renal pedicle is reached. The renal pedicle will then be isolated while maintaining traction on the kidney, and peri-renal fat, and ligated using Weck® clips. A second peripheral blood sample will be collected at the time of specimen extraction. A third and fourth peripheral blood samples will be collected at post-operative days 1 and 30, respectively, to study CTC post-op kinetics. All samples will collect 7.5 mL of peripheral blood.

Patients presenting with hypofunctioning kidneys with indication for total nephrectomy will be used as controls. Total nephrectomy patients will undergo the randomization protocol, in a control arm.

The CTCs will be isolated from peripheral blood samples using a microfluidics size-based CTC capture device - Ruby™. Whole blood samples will be injected into the devices at an 80 µL/min flow rate. The CTCs captured on the devices will then be stained with antibodies to 4',6-diamidino-2-phenylindole (DAPI) to identify cell nuclei, cluster of differentiation antigen 45 (CD45) to identify leukocytes, cytokeratin 8/18 to identify epithelial CTCs, and vimentin to identify mesenchymal CTCs or CTCs which have undergone epithelial-to-mesenchymal transition. Blood samples will be processed no more than 30 minutes after collection.

ELIGIBILITY:
Inclusion Criteria:

* Renal mass on renal imaging compatible with kidney cancer
* Indication for laparoscopic radical nephrectomy

Exclusion Criteria:

* History of other cancer (carcinoma)
* Previous systemic therapy for renal cell carcinoma
* human immunodeficiency virus (HIV) positive
* Hepatitis C virus (HCV) positive
* hepatitis B virus (HBV) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Circulating tumor cell count - intra-operative | Intra-operative
  CTC count in peripheral blood after tumor specimen extraction
Circulating tumor cell count - D1 | Post-operative day 1
  CTC count in peripheral blood at post-operative day 1
Circulating tumor cell count - D30 | Post-operative day 30
  CTC count in peripheral blood at post-operative day 30

SECONDARY OUTCOMES:
Overall survival | 3 year
  Overall survival
Disease free survival | 3 year
  Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Tito P Leitão, MD, Principal Investigator — Faculdade de Medicina da Universidade de Lisboa
Locations (1):
- Urology Department - Hospital de Santa Maria, Lisbon, Lisbon District, Portugal